CLINICAL TRIAL: NCT05692947
Title: The Validity of CORE Sensor in Heat Training for Male and Female Endurance Athletes
Acronym: CORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000607
Record Dates: First submitted 2022-09-12; First posted 2023-01-20 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Temperature Change, Body
Keywords: Exercise; Heat acclimation; Core temperature; Heat loading; Heat stress; Thermoregulation
MeSH Terms: conditions — Body Temperature Changes; Motor Activity; Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: Each athlete will be asked to exercise for 45 minutes in a hot/dry condition (38 degrees Celsius and 10-20% relative humidity) and a hot/humid condition (28 degrees Celsius and 80-100% relative humidity). Experimental sessions will occur at least seven days apart and participants will be randomly assigned to which condition they experience first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Hot/Dry (Experimental): Core body temperature, skin temperature, heart rate, and heat perceptions will be collected from elite athletes while running or cycling for 45 minutes in the heat at low humidity (38 degrees Celsius with 10-20% relative humidity).
  Interventions: Device: Core body temperature device
- Hot/Humid (Experimental): Core body temperature, skin temperature, heart rate, and heat perceptions will be collected from elite athletes while running or cycling for 45 minutes in the heat at high humidity (28 degrees Celsius with 80-100% relative humidity).
  Interventions: Device: Core body temperature device

INTERVENTIONS:
Device: Core body temperature device — This study is to verify the claims of CORE™ body temperature system to estimate core body temperature from skin temperature and heart rate during exercise under varying environmental conditions. Subjects will ingest a temperature sensing pill and be outfitted with skin temperature sensors, a chest strap heart rate monitor, and the CORE and CaleraResearch devices. Athletes will run or cycle in hot/dry and hot/humid conditions for 45 minutes at an absolute workload of 60% VO2 Max/Peak.
  Other Names: CORE™; CaleraResearch™

SUMMARY:
This study is investigating the efficacy of CORE™ devices in calculating core body temperature in athletes under varying environmental conditions.

DETAILED DESCRIPTION:
As athletes exercise, their core body temperature rises, which can affect their performance. Additionally, repeated mild to moderate heat stress, heat acclimation, can be used to improve exercise tolerance and performance. Thus, an athlete can gain performance benefits through monitoring their heat loading while training. The aim of this study is to compare the CORE™ body temperatures recorded during exercise in two different environmental conditions in which the investigators will get a separation of core temperature and skin temperature. The investigators will accomplish this by recruiting trained and elite athletes, ages 18-59, to participate in two exercise sessions in the heat at low (10-20%) and high (80-100%) relative humidity. The investigators will compare the CORE™ temperature estimates against an FDA approved ingestible temperature monitoring device to assess the accuracy of the CORE™ devices.

ELIGIBILITY:
Inclusion Criteria:

* Highly trained or elite athlete
* Nonsmokers
* Able to read and speak English
* No underlying cardiovascular limitations

Exclusion Criteria:

* Currently or previously a habitual smoker (nicotine/cannabis)
* Pregnant, breast feeding, trying to conceive, undergoing treatment to increase sperm count
* Those taking medications that affect cardiovascular function, with the exception of oral contraceptives
* History of stroke, clotting disorders or venous thrombosis
* A history of heat illness or heat injury
* History of obstructive diseases of the gastrointestinal tract including diverticulosis, diverticulitis, inflammatory bowel disease, peptic ulcer disease, Chron's disease, ulcerative colitis, or previous GI surgery

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Ability to accurately estimate core body temperature | 30 minutes
  The CORE and CaleraResearch devices estimate core body temperature using single-site skin temperature and heartrate as data inputs for their proprietary algorithm. This calculated temperature will be assessed against actual core body temperature, measured with an FDA approved, ingestible, temperature-sensing telemetry pill.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher T Minson, PhD, Principal Investigator — University of Oregon
Locations (1):
- Bowerman Sports Science Center at the University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT05692947/ICF_000.pdf